CLINICAL TRIAL: NCT05696600
Title: "Impact of Supracrestal Tissue Attachment Dimension on the Outcome of Scaling and Root Planing and Open Flap Debridement Procedure in Patients With Stage II and Stage III Periodontitis in Thin Versus Thick Periodontal Phenotype: A Comparative Interventional Study"
Brief Title: Impact of Supracrestal Tissue Attachment Dimension on Outcome of Scaling and Root Planing and Open Flap Debridement Procedure in Different Periodontal Phenotypes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAKSHIPERIO
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thick periodontal phenotype (Experimental): Scaling and root planing and open flap debridement in patients with stage II and stage III periodontitis
  Interventions: Procedure: Scaling and root planing and open flap debridement
- Thin periodontal phenotype (Active Comparator): Scaling and root planing and open flap debridement in patients with stage II and stage III periodontitis
  Interventions: Procedure: Scaling and root planing and open flap debridement

INTERVENTIONS:
Procedure: Scaling and root planing and open flap debridement — Scaling and root planing involves removal of plaque and calculus.
  Open Flap debridement involves reflection of full thickness mucoperiosteal flap, thorough debridement of the surgical site and approximation and suturing of the flap at the original position.

SUMMARY:
The existence of supracrestal tissue attachment (SCTA) is fundamental for adhesion of the junctional epithelium and insertion of the connective fibers to the dental structure, besides functioning as a barrier against microbial entry in the periodontium. Wide variation in SCTA dimension have been reported in patients with and without periodontitis. If the physiologic dimension of SCTA is violated then it may lead to inflammation in periodontium. Influence of dimension of SCTA on scaling and root planning and open flap debridement procedure has not been investigated till date. Thus the aim of study is to assess the influence of SCTA dimension on the outcome of scaling and root planning followed by open flap debridement in patients with stage 2 and stage 3 periodontitis and also to estimate the SCTA dimension in thick versus thin periodontal phenotype.

DETAILED DESCRIPTION:
Periodontitis is defined as an inflammatory disease of supporting tissues of teeth caused by specific microorganisms or groups of specific microorganisms, resulting in progressive destruction of the periodontal ligament and alveolar bone with periodontal pocket formation, gingival recession or both 1. Its severe form affects 11% of the population worldwide 2. Periodontitis influence oral health related quality of life (OHRQoL) and thus is a major public health problem3. Treatment of periodontal disease includes non-surgical and surgical procedures. Reduction in pocket depth and gain in clinical attachment level are usually considered as successful outcomes of periodontal therapy. While Non-surgical therapy is effective in shallow pockets, significant gain of clinical attachment is usually observed in deep pockets after surgical therapy 4.

There are various surgical procedures for the management of periodontal pocket which include curettage, gingivectomy, periodontal flap surgery and guided tissue regeneration. Among these, periodontal flap surgery is used widely. The primary objective of periodontal flap surgery is to obtain access for root instrumentation so that plaque can be removed and the secondary objective is pocket reduction via soft and hard tissue resection to facilitate home care5. Neumann was the pioneer of periodontal flap6 surgery then Widman described the different incision technique for periodontal flap in 1966. A modification of Widman flap was described by Ramfjord and Nissle in 19747. This modification includes initial incision which is parallel to the long axis to the tooth and a second crevicular incision which surrounds the neck of teeth. Advantages of modified Widman flap surgery are that it conserves bone and there is optimal root coverage which is esthetically acceptable and also permits oral hygiene. It also results in more pocket closure and more bone regeneration. But one of the major disadvantage of modified Widman flap procedure is unfavourable interproximal architecture immediately after removal of dressing7.

With time it has been seen that outcomes of surgical periodontal therapy is effectively influenced by various factors such as pocket depth, severity of gingival inflammation, marginal alveolar bone, systemic diseases and smoking8-10. As per the literature available these factors need to be further explored. Biologic width, which is now known as supracrestal tissue attachment (SCTA) is described as a variable entity comprising of junctional epithelium and connective tissue attachment coronal to the alveolar crest11. A landmark histologic study by Gargiulo et al which was done on human autopsy specimens has given an average of 2.04 mm for this entity12, though a study by Vacek et al stated that it may range from 0.75 mm to as large as 4 mm in a healthy periodontium13. But these studies did not tell about the clinical significance of BW and then Inger et al were the first to describe the clinical significance of biological width in dentistry. Another human histometric study has demonstrated mean measurement of supracrestal tissue as 2.75+/-0.59mm. however these studies were only conducted on healthy periodontium14. Only a few studies have attempted to assess the dimensions of SCTA in periodontal disease. According to a study by Novak et al, average clinical biologic width in case of severe, generalized, chronic periodontitis was observed to be nearly twice as previously reported for histological width which was 2.04mm (1.94 -1.97mm). In this study 44% of all measured sites were had PD and CAL less than equal to 3mm. Its observations suggested that even in the presence of a severe, generalized, horizontal pattern of alveolar bone loss, nearly half of the clinical sites in the mouth showed minimal clinical signs of disease but extensive radiographic evidence of alveolar bone loss15. One of the study by Abullais et al suggest that clinical and radiographic findings of the SCTA showed a significant difference in patients with periodontitis16. Various clinical and experimental studies are available in the literature about the effect of periodontal surgical procedure on healing and regeneration of SCTA but there is no study in the literature which demonstrate the effect of SCTA on scaling and root planning and open flap debridement. Thus, the aim of this study is to evaluate the impact of supracrestal tissue attachment dimension on the outcomes of scaling and root planing followed by open flap debridement in patients with stage 2 and stage 3 periodontitis between thick versus thin periodontal phenotypes.

MATERIALS AND METHODOLOGY

SETTINGS: The present prospective clinical trial will be conducted in the Department of Periodontics, Post Graduate Institute of Dental Sciences, Rohtak STUDY DESIGN: Interventional study TIME FRAME: 12-14 months SAMPLE SIZE Sample size determination was done by using G power software. Results of a previous study by Gumber et al. taking changes in clinical attachment gain as the clinical outcome at the end of 6 months between thick and thin PP was used to compute the effect size, taking power as 80% and α as 0.05. Sample of 18 patients per group was calculated as the minimum sample size for the study. Considering 30% patient attrition, a total of 24 patients will be recruited per group.

METHOD OF RECRUITMENT:

Patients will be recruited from out patient clinic of Department of Periodontics, PGIDS, Rohtak after screening based on given inclusion and exclusion criteria.

RANDOMIZATION & ALLOCATION CONCEALMENT-Not applicable BLINDING/MASKING-single blind INTERVENTION All the participants will undergo phase-I therapy with a combination of hand scalers and curettes (Hu Friedy) and ultrasonic scaler (EMS Piezon,250, Switzerland). Oral hygiene instructions will be imparted and will be reinforced at each appointment.

After a period of 6 weeks of scaling and root planing, patients having residual probing depth of ≥ 5 mm at ≥ 4 sites along ≥ 2 maxillary or mandibular incisors teeth will be recalled for open flap debridement. Patients will be recalled at the end of 3 months and 6 months for recording of parameters.

METHODOLOGY:

Patients fulfilling the eligibility criteria will be enrolled in the study after obtaining the informed consent. Periodontal parameters will be assessed which include Plaque index (PI), Gingival index (GI), clinical attachment level (CAL) , periodontal pocket depth (PPD), bleeding on probing (BOP), Periodontal phenotype (PP), keratinized tissue width (KTW) and supracrestal tissue attachment (SCTA).

KTW will be evaluated before supracrestal tissue attachment (SCTA) measurement and SCTA will be measured under local anesthesia.

The transgingival probing depth will be measured till the alveolar crest (from the free gingival margin to the alveolar crest under LA). SCTA will be obtained after subtracting the probing depth (free gingival margin to base of the periodontal pocket) from supracrestal gingiva.

Evaluation of PP will be done after completion of Phase I therapy using probe transparency method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with generalised stage II or stage III periodontitis
2. Maxillary or mandibular incisors having same periodontal phenotype

Exclusion Criteria:

1. Patient with systemic diseases like uncontrolled diabetes, hypertension, bleeding disorders, coronary artery disease etc.
2. Malaligned teeth
3. Patient having undergone any periodontal therapy within one year
4. Pregnant and lactating females
5. Patient on antibiotic therapy in the past one month

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
CLINICAL ATTACHMENT LEVEL (CAL) | 6 MONTHS
  Clinical Attachment Level will be measured as the distance between the base of the clinical pocket and the cemento-enamel junction(CEJ).Measurements will be made at 6 sites of involved tooth- mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto- lingual using UNC-15 probe.
BLEEDING ON PROBING (BOP) | 6 MONTHS
  BOP will be recorded as 1 (present) if it occurred within 15 sec of probing and 0 (absent) if no bleeding occurred. It will be calculated in %. After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100. It will be designed as % sites with bleeding on probing.
PROBING POCKET DEPTH (PPD) | 6 MONTHS
  Probing pocket depth will be measured as the distance from the gingival margin to the base of the clinical pocket. The probing depth measurements will be assessed using a calibrated manual periodontal probe (PCP-UNC 15 Hu-Friedy, Chicago, IL, USA). The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of involved tooth - mesio-buccal, mid-buccal, disto-buccal, mesio- lingual, mid-lingual, disto-lingual. Measurements will be rounded to the nearest whole millimetre.

CONTACTS AND LOCATIONS:
Overall Officials: SAKSHI VERMA, BDS, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No